CLINICAL TRIAL: NCT02729298
Title: A Phase 1a / 1b, First-in-human, Open-label, Dose-escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral TP-0903 Administered Daily for 21 Days to Patients With Advanced Solid Tumors
Brief Title: First-in-human Study of Oral TP-0903 (a Novel Inhibitor of AXL Kinase) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP-0903-101
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumors; EGFR Positive Non-small Cell Lung Cancer; Colorectal Carcinoma; Recurrent Ovarian Carcinoma; BRAF-Mutated Melanoma
Keywords: Tolero; Phase 1a / 1b; First in human; Solid Tumors with immunotherapy progression; AXL inhibitor; Advanced Malignancy; Cancer; EGFR+ NSCLC with progression on ≤2 lines of oral TKIs; BRAF-Mutated CRC; KRAS-Mutated CRC; NRAS-Mutated CRC; Persistent/Recurrent Ovarian Cancer; BRAF-Mutated Melanoma with immunotherapy progression
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Neoplasms | interventions — dubermatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Advanced Solid Tumors (Experimental): Phase 1a Single daily dose of TP-0903 by oral administration on Days 1-21 of a 28 day cycle
  AND
  Phase 1b - Upon confirmation of MTD, will receive single oral daily doses of a flat dose of TP-0903 based on the average of the dose administered in the MTD expansion safety cohort on Days 1-21 of each 28 day cycle.
  Interventions: Drug: TP-0903
- EGFR+ NSCLC (Experimental): Phase 1b - Upon confirmation of MTD, will receive single oral daily doses of a flat dose of TP-0903 based on the average of the dose administered in the MTD expansion safety cohort on Days 1-21 of each 28 day cycle.
  Interventions: Drug: TP-0903
- BRAF-, KRAS-, or NRAS-Mutated CRC (Experimental): Phase 1b - Upon confirmation of MTD, will receive single oral daily doses of a flat dose of TP-0903 based on the average of the dose administered in the MTD expansion safety cohort on Days 1-21 of each 28 day cycle.
  Interventions: Drug: TP-0903
- Persistent/Recurrent Ovarian Cancer (Experimental): Phase 1b - Upon confirmation of MTD, will receive single oral daily doses of a flat dose of TP-0903 based on the average of the dose administered in the MTD expansion safety cohort on Days 1-21 of each 28 day cycle.
  Interventions: Drug: TP-0903
- BRAF-Mutated Melanoma (Experimental): Phase 1b - Upon confirmation of MTD, will receive single oral daily doses of a flat dose of TP-0903 based on the average of the dose administered in the MTD expansion safety cohort on Days 1-21 of each 28 day cycle.
  Interventions: Drug: TP-0903

INTERVENTIONS:
Drug: TP-0903 — Novel oral inhibitor that targets AXL kinase and reverses the mesenchymal phenotype associated with advanced cancers

SUMMARY:
TP-0903 is a novel oral inhibitor that targets AXL kinase and reverses the mesenchymal phenotype associated with advanced cancers. Preclinical studies have shown promising antitumor activity of TP-0903 as a single agent against a variety of tumor types in both in vitro and in vivo studies.

This first-in-human Phase 1a study is conducted to identify the maximum tolerated dose (MTD) of TP-0903 administered orally to patients with advanced solid tumors and to identify the safety profile and Recommended Phase 2 Dose (RP2D) of TP-0903. Once the MTD has been established, additional patients with specific tumor types (advanced solid tumors that have progressed after achieving a best documented response of at least stable disease (ie, SD, PR, or CR documented per iRECIST following at least 2 cycles (8 weeks) of immunotherapy, EGFR+ Non Small Cell Lung Cancer [NSCLC] and have demonstrated recent progression following a best documented response of at least stable disease (ie, SD, PR, or CR documented per RECIST v1.1 on ≤2 lines of oral TKIs (Prior chemotherapy ± immunotherapy is allowed as long as the patient is clearly demonstrating current progression on an EGFR TKI.), BRAF-, KRAS-, or NRAS-mutated Colorectal Carcinoma [CRC] for whom there is no standard therapy remaining, persistent/recurrent Ovarian Cancer who would be platinum refractory/ resistant and have had any number of lines of prior therapy, and BRAF-mutated Melanoma that has not responded to immunotherapy or a combination BRAF/MEK inhibitor) will be enrolled at the MTD in the Phase 1b study. Data collected from patients enrolled in each of these additional cohorts will be used for to confirm safety, explore potential biomarkers, and evaluate potential signals of activity when TP-0903 is administered to specific groups of heavily pretreated patients or given in combination with immunotherapy or a tyrosine kinase inhibitor (TKI).

The study will investigate the safety, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity profiles.

DETAILED DESCRIPTION:
This is a phase 1a / 1b, first-in-human, open-label, dose-escalation, safety, pharmacokinetics, and pharmacodynamic study of TP-0903 administered once daily for the first 21 out of 28 days.

There are 2 phases in this study. In Phase 1a (dose escalation), sequential cohorts of three (3) patients will be treated with escalated doses until the MTD is established. In the absence of dose-limiting toxicities (DLTs), the dose will be increased using a modified Fibonacci dose escalation scheme.

Once the MTD has been established, dosing will change from BSA-dependent to a flat dose based on the average of the dose administered in the MTD expansion safety cohort. Once the MTD has been established, in Ph 1b (expansion), 5 additional cohorts of up to 20 patients each with specific tumor types (up to 100 additional patients total) may be enrolled at the MTD dose level to confirm safety, explore potential biomarkers, and evaluate potential signals of activity when TP-0903 is administered to specific groups of heavily pretreated patients or given in combination with immunotherapy or a tyrosine kinase inhibitor (TKI). Ten patients in each of these 5 Expansion Cohorts will be required to consent to undergo pre- and post-dose tumor biopsies. All patients who undergo these biopsies will comprise the 'Biopsy Cohorts' (Phase 1b).

Patients who successfully complete a 4-week treatment cycle without evidence of significant treatment-related toxicity or progressive disease will be permitted to continue to receive treatment with the same dose and dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in the study, patients must meet all of the following inclusion criteria:

1. Patients enrolled in the Phase 1a study must:

   1. Have a histologically confirmed diagnosis of advanced metastatic or progressive solid tumor
   2. Be refractory to, or intolerant of, established therapy known to provide clinical benefit for their condition
2. Patients enrolled in the Phase 1b study must meet criteria for one of the following tumor types:

   1. Have tumors that have progressed after achieving a best documented response of at least stable disease (ie, SD, PR, or CR documented per iRECIST following at least 2 cycles (8 weeks) of immunotherapy and are felt to be appropriate for this type of treatment*
   2. Have EGFR+ NSCLC and have demonstrated recent progression following a best documented response of at least stable disease (ie, SD, PR, or CR documented per per RECIST v1.1 on ≤2 lines of oral TKIs and are felt to be appropriate for this type of treatment* Prior chemotherapy ± immunotherapy is allowed as long as the patient is clearly demonstrating current progression on an EGFR TKI.
   3. Have BRAF-, KRAS-, or NRAS-mutated CRC for whom there is no standard therapy remaining
   4. Have persistent/recurrent ovarian cancer who would be platinum refractory/ resistant and have had any number of lines of prior therapy
   5. Have BRAF-mutated melanoma that has not responded to immunotherapy or a combination BRAF/MEK inhibitor
3. Have one or more tumors measurable or evaluable as outlined by modified RECIST v1.1 or iRECIST
4. Have an Eastern Cooperative Oncology Group (ECOG) (World Health Organization [WHO]) performance of ≤1
5. Have a life expectancy ≥3 months
6. Be ≥18 years of age
7. Have a negative pregnancy test (if female of childbearing potential)
8. Have acceptable liver function:

   1. Bilirubin ≤1.5x upper limit of normal (ULN)

      *Patients receiving immunotherapy should have a bilirubin level <3.0x ULN.
   2. Aspartate aminotransferase (AST/SGOT), alanine aminotransferase (ALT/SGPT) and alkaline phosphatase ≤2.5x upper limit of normal (ULN)

      * If liver metastases are present, then ≤5x ULN is allowed.
      * Patients receiving immunotherapy should have AST and ALT levels <5.0x ULN.
9. Have acceptable renal function:

   a. Calculated creatinine clearance ≥30 mL/min
10. Have acceptable hematologic status:

    1. Granulocyte ≥1500 cells/mm3
    2. Platelet count ≥100,000 (plt/mm3)
    3. Hemoglobin ≥9 g/dL
11. Have no clinically significant abnormalities on urinalysis
12. Have acceptable coagulation status:

    1. Prothrombin time (PT) within 1.5x normal limits
    2. Activated partial thromboplastin time (aPTT) within 1.5x normal limits
13. Be nonfertile or agree to use an adequate method of contraception. Sexually active patients and their partners must use an effective method of contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation and for at least 30 days after the last study drug dose (see Section 4.6.3). Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
14. Have read and signed the IRB-approved informed consent form prior to any study related procedure. (In the event that the patient is re-screened for study participation or a protocol amendment alters the care of an ongoing patient, a new informed consent form must be signed.)
15. Patients enrolled in each of the five Expansion Cohorts must be willing to consider pre-study and on-study biopsies, if safe and medically feasible, as determined by local interventional radiology (3 to 5 core samples requested at each biopsy timepoint)

Patients meeting any one of these exclusion criteria will be prohibited from participating in this study:

1. Have New York Heart Association (NYHA) Class III or IV, cardiac disease, myocardial infarction within the past 6 months prior to Day 1, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG) or during Cardiac Stress Testing within 14 days prior to Day 1 (Appendix C)
2. Have a corrected QT interval (QTcF, Fridericia's method) of >450 msec in men and >470 msec in women
3. Have a seizure disorders requiring anticonvulsant therapy
4. Presence of symptomatic central nervous system metastatic disease or disease that requires local therapy such as radiotherapy, surgery, or increasing dose of steroids within 2 weeks prior to Day 1
5. Have severe chronic obstructive pulmonary disease with hypoxemia (defined as resting O2 saturation of ≤88% breathing room air)
6. Have undergone major surgery, other than diagnostic surgery, within 2 weeks prior to Day 1
7. Have active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
8. Are pregnant or nursing
9. Received treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within 28 days or 5 half lives, whichever occurs first, prior to study entry (6 weeks for nitrosoureas or Mitomycin C)

   a. This exclusion criterion is not applicable for patients with EGFR+ NSCLC or immunotherapy-resistant tumors who are enrolled in expansion cohorts at the MTD.
10. Are unwilling or unable to comply with procedures required in this protocol
11. Have known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C. Patients with history of chronic hepatitis that is currently not active are eligible
12. Have a serious nonmalignant disease (eg, hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
13. Are currently receiving any other investigational agent
14. Have exhibited allergic reactions to a similar structural compound, biological agent, or formulation
15. Have undergone significant surgery to the gastrointestinal tract that could impair absorption or that could result in short bowel syndrome with diarrhea due to malabsorption
16. Have a history of severe adverse reaction (eg, hypersensitivity reaction, anaphylaxis) to sulfonamides
17. Patients scheduled to receive immunotherapy or TKI regimens plus TP-0903 must not be currently taking high-dose steroids (ie, physiologic dose approximately equivalent to 15 mg/day of prednisone)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) and treatment emergent adverse events | Cycle 1 (Day 1 through Day 28)
  A DLT is defined as any one of the following events observed within Cycle 1:
  Grade 3 or greater febrile neutropenia, Grade 4 ANC for 7 or greater consecutive days, Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with clinically significant bleeding or that requires a platelet transfusion, Grade 3 or 4 non-hematologic AEs including nausea, vomiting, diarrhea, and electrolyte imbalances persisting for more than 48 hours despite optimal medical management, dosing delays of 2 weeks or greater due to treatment emergent adverse events or related severe laboratory test values

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from zero to infinity [AUC(0-inf)] of oral TP-0903 | Cycles 1 and 2 (Day 1 through 23)
  Derived PK parameters by non-compartment analysis on Cycle 1.
Area under the plasma concentration-time curve from zero to last measured time point [AUC(0-last)] of oral TP-0903 | Cycles 1 and 2 (Day 1 through 23)
  Derived PK parameters by non-compartment analysis on Cycle 1
Peak plasma concentration (Cmax) of oral TP-0903 | Cycles 1 and 2 (Day 1 through 23)
  Derived PK parameters by non-compartment analysis on Cycle 1.
Activity of TP-0903 on predictive biomarkers | End of every cycle (each cycle is 28 days) and End of Study (within 14 days of the last dose of study drug or within 14 days of the decision to discontinue study treatment)
  Assess biomarkers in tumor tissue, PBMCs, plasma and serum. The pharmacodynamic relationships of TP-0903 exposure with exploratory biomarkers will be quantified using the Spearman rank correlation statistic.
Objective response rate using RECIST v1.1 and iRECIST | End of every cycle (each cycle is 28 days) and End of Study (within 14 days of the last dose of study drug or within 14 days of the decision to discontinue study treatment)
  Baseline tumor assessment will be performed at screening and repeated at Cycle 2 and every even cycle thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Anthony, DO, Study Director — Sumitomo Pharma America, Inc.
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Colorado Denver, Denver, Colorado
  - US Oncology - Rocky Mountain Cancer Centers, LLP (RMCC), Denver, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - University of Kansas Cancer Center, Fairway, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - US Oncology - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - US Oncology - Texas Oncology Austin, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - US Oncology - Texas Oncology - Fort Worth, Fort Worth, Texas
  - University of Texas Science Center at San Antonio (UTHSCSA), San Antonio, Texas
  - US Oncology - Texas Oncology - Tyler, Tyler, Texas
  - US Oncology - Virginia Cancer Specialists (VCS), Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No